CLINICAL TRIAL: NCT00006397
Title: A Study of the Combination of Indinavir, Ritonavir, Enteric-Coated ddI and d4T In Nucleoside and Non-Nucleoside Reverse Transcriptase Inhibitor Experienced Patients: An Open-Label Study Investigating Differences Between Women and Men
Brief Title: Differences Between Women and Men Taking a Combination of Indinavir, Ritonavir, Enteric-Coated Didanosine, and Stavudine Who Previously Took Anti-HIV Drugs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PPD Development, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 312A; BMS 2000
Record Dates: First submitted 2000-10-10; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Sex Factors; Ritonavir; Indinavir; Dosage Forms; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Stavudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see how safe and effective it is to give multi-drug treatment with indinavir (IDV) plus ritonavir (RTV) plus enteric-coated didanosine (ddI) plus stavudine (d4T) and if there are differences in responses between men and women.

DETAILED DESCRIPTION:
Patients are enrolled in balanced numbers based on gender and stratified by viral load (less than or equal to 10,000, 10,000 to 100,000, or more than 100,000 copies/ml). Prior to therapy, a peer-based patient education intervention is presented. Patients receive a combination of IDV, RTV, enteric-coated ddI, and d4T. Responses to this multi-agent antiretroviral drug regimen are explored based on sex differences. A pharmacokinetic sub-study, balanced so that half of patients are male and half are female, is performed on IDV and RTV for 20 to 25 of the patients. About 20 females are examined for study-drug effects on gonadotropic hormone levels.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have viral load (amount of HIV in the blood) greater than 500 copies/ml.
* Have received anti-HIV treatment previously with an NNRTI plus an NRTI combination or only NRTIs for greater than 8 weeks and, if not currently on treatment, have been off treatment for 12 weeks or less.
* Failed to keep their viral load low during previous anti-HIV treatment.
* Are at least 18 years of age.
* Agree to use an effective barrier method of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have used a protease inhibitor for more than 14 days.
* Have used ddI or d4T for more than 30 days.
* Are pregnant or breast-feeding.
* Have an opportunistic (AIDS-related) infection requiring treatment at the time of enrollment.
* Have, or appear to have, peripheral neuropathy (a painful condition affecting the nervous system) at the time of screening.
* Are at risk for, or have had, pancreatitis (disease of the pancreas).
* Have difficulty absorbing medications.
* Have a cancer, other than Kaposi's sarcoma, that may require systemic treatment.
* Have any medical condition or treatment that may cause a rise in viral load.
* Have any other condition or previous treatment that would interfere with the study.
* Are unable to take drugs by mouth.
* Are receiving or have received recently any of the following drugs: terfenadine, astemizole, cisapride, triazolam, midazolam, ergot alkaloids, amiodarone, bepridil, flecainide, propafenone, quinidine, pimozide, rifampin, and intravenous (IV) pentamidine.
* Are receiving vincristine, thalidomide, foscarnet, or cisplatin or other medications that may cause nerve damage.
* Have received any experimental drug within 30 days prior to treatment.
* Are receiving treatment with testosterone, anabolic steroids, growth hormone, or megestrol acetate, except for certain hormonal problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - East Bay AIDS Ctr, Berkeley, California
  - Univ of Southern California, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - North Broward Hosp District / HIV Clinical Research, Fort Lauderdale, Florida
  - Saint Josephs Comprehensive Research Institute, Tampa, Florida
  - Louisiana State Univ Med Ctr / HIV Outpatient Clinic, New Orleans, Louisiana
  - JSI Research and Training Institute, Boston, Massachusetts
  - Univ of Med & Dentistry of New Jersey, Newark, New Jersey
  - Beth Israel Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Vanderbilt Univ School of Medicine, Nashville, Tennessee
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
- Puerto Rico (2):
  - Ponce Univ Hosp, Ponce
  - Univ of Puerto Rico School of Med, Rio Piedras